CLINICAL TRIAL: NCT00240422
Title: A Prospective, Randomized, Double-blind, Double-dummy, Forced Titration, Parallel Group Comparison, Multicenter Trial to Compare the Effects of Either Telmisartan (40-80 mg p.o. Once Daily) or Ramipril (5-10 mg p.o. Once Daily) on Renal Endothelial Dysfunction in Hypertensive Patients With Type 2 Diabetes
Brief Title: Trial to Compare the Effects of Either Telmisartan (40-80 mg PO Once Daily) or Ramipril (5-10 mg PO Once Daily) on Renal Endothelial Dysfunction in Hypertensive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.398
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Telmisartan; Ramipril

INTERVENTIONS:
Drug: Telmisartan
Drug: Ramipril

SUMMARY:
The primary objective is to evaluate the effect of 9 weeks treatment with either telmisartan or ramipril on NO bioavailability in the renal vasculature, measured as renal plasma flow (RPF) in response to NG-monomethyl-L-arginine (LNMMA) infusion.

DETAILED DESCRIPTION:
This study was designed as a randomised, double-blind, double-dummy, parallel group in hypertensive patients with type 2 diabetes and normo- or microalbuminuria over a treatment period of 9 weeks.

After a 4 week Run-in period, patients will be randomised to one of the treatment groups and receive either Telmisartan 40 - 80 mg or Ramipril 5 - 10 mg. The treatment regimen is a forced titration with the lower dose given for 3 weeks and the higher dose given for the rest of the treatment period summing up to 9 weeks of treatment. During the treatment period, 3 visits to the investigator will be scheduled in order to control blood pressure, renal function parameters and safety. In addition, parameters of endothelial function in the renal vasculature, based on a nephrological clearance investigation and a provocation with L-NMMA will be measured at baseline and after 9 weeks of treatment.

Study Hypothesis:

Due to the exploratory nature of the trial, the primary objective to evaluate the effect on RPF in response to L-NMMA infusion at baseline and after 9 weeks of therapy with either telmisartan 80 mg or ramipril 10 mg was not planned to be addressed by a test of prespecified hypotheses.

Comparison(s):

The change in RPF from baseline (Visit 4) to the end of treatment (Visit 7) in response to L-NMMA infusion was to be calculated as the change from the pre L-NMMA infusion (S1) to the end of the L-NMMA infusion (S2). A comparison of treatment groups was to be made using an analysis of covariance (ANCOVA) with pooled centre and treatment included as main effects and RPF (in response to L NMMA infusion) at baseline as a covariate. The treatment group difference, adjusted for the other factors in the model, was to be presented with a corresponding 95% confidence interval (CI) and a test of statistical significance. The model was also to be used to provide analysis results for the within treatment group changes.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients aged 30-80 years with type 2 diabetes, normo- or microalbuminuria, GFR > 80 mL/min (Cockroft-Gault)

Exclusion Criteria: None

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2003-02; Study Completion 2004-07

PRIMARY OUTCOMES:
Change from baseline of renal plasma flow (RPF) in response to L-NMMA infusion at the end of treatment. | 9 weeks

SECONDARY OUTCOMES:
Change from baseline of glomerular filtration rate (GFR) in response to L-NMMA infusion at the end of treatment | 9 weeks
Change from baseline of filtration fraction (FF) in response to L-NMMA infusion at the end of treatment. | 9 weeks
Change from baseline of renal vascular resistance (RVR) in response to L-NMMA infusion at the end of treatment. | 9 weeks
Change from baseline of RPF in response to L-arginine infusion at the end of treatment. | 9 weeks
Change from baseline of GFR in response to L-arginine infusion at the end of treatment | 9 weeks
Change from baseline of FF in response to L-arginine infusion at the end of treatment. | 9 weeks
Change from baseline of RVR in response to L-arginine infusion at the end of treatment. | 9 weeks
Change from baseline of mean arterial pressure (MAP) and pulse rate (PR) in response to L-NMMA infusion at the end of treatment. | 9 weeks
Change from baseline of MAP and PR in response to L-arginine infusion at the end of treatment. | 9 weeks
Change from baseline of the laboratory parameters angiotensin II (ANG II), aldosterone, asymmetrical dimethylarginine (ADMA), L-arginine, urinary nitrate/nitrite (UNOx), and urinary albumin excretion at the end of treatment | 9 weeks
Change from baseline of the pre-L-NMMA RPF at the end of treatment | 9 weeks
Change from baseline of the pre-L-NMMA GFR at the end of treatment | 9 weeks
Change from baseline of the pre-L-NMMA FF at the end of treatment. | 9 weeks
Change from baseline of the pre-L-NMMA RVR at the end of treatment. | 9 weeks
Change from baseline of the urinary excretion parameters creatinine, sodium, potassium, and urea at the end of treatment. | 9 weeks
Blood pressure response and control at the end of treatment | 9 weeks
Change from baseline of central blood pressure and augmentation index (by pulse wave analysis) at the end of treatment. | 9 weeks
Change from baseline of RPF in response to Vitamin C infusion at the end of treatment | 9 weeks
Change from baseline of GFR in response to Vitamin C infusion at the end of treatment | 9 weeks
Change from baseline of FF in response to Vitamin C infusion at the end of treatment. | 9 weeks
Change from baseline of RVR in response to Vitamin C infusion at the end of treatment. | 9 weeks
Change from baseline of MAP and PR in response to Vitamin C infusion at the end of treatment. | 9 weeks
Incidence of adverse events | week -2 and 9 weeks
Changes from base line in routine laboratory data at the end of the study | 9 weeks
Changes in vital signs | 9 weeks
Changes from screening in physical examination at the end of the study | - 4 weeks and 9 weeks
Changes from screening in ECG at the end of the study | - 4 weeks and 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (6):
- France (2):
  - Boehringer Ingelheim Investigational Site, Lyon
  - Boehringer Ingelheim Investigational Site, Montpellier
- Germany (3):
  - Friedrich-Alexander-Universität, Erlangen
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Universität Erlangen-Nürnberg, Nuremberg
- Edificio de Medicina Comunitaria, Madrid, Spain

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786